CLINICAL TRIAL: NCT01948830
Title: A 12-month, Phase 3b, Randomized, Visual Acuity Assessor-masked, Multicenter Study Assessing the Efficacy and Safety of Ranibizumab 0.5mg in Treat and Extend Regimen Compared to Monthly Regimen, in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Randomized Study for Efficacy and Safety of Ranibizumab 0.5mg in Treat-extend and Monthly Regimens in Patients With nAMD
Acronym: TREND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CRFB002A2411; 2013-002626-23 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Age-related Macular Degeneration; Choroidal Neovascularization
Keywords: Ranibizumab, Lucentis, choroidal neovascularization, age-related macular degeneration, treat and extend regimen
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I ranibizumab 0.5 mg monthly (Active Comparator): Ranibizumab 0.5 mg/0.05 mL (Monthly regimen) up to month 11
  Interventions: Drug: Ranibizumab 0.5mg
- Group II ranibizumab 0.5 mg TER (Active Comparator): Ranibizumab 0.5 mg/0.05 mL (TER) treat and Extend regimen up to month 11
  Interventions: Drug: Ranibizumab 0.5mg

INTERVENTIONS:
Drug: Ranibizumab 0.5mg — 0.5 mg ranibizumab (intravitreal injections) prefilled syringe)
  Other Names: Lucentis
  Arms: Group I ranibizumab 0.5 mg monthly
Drug: Ranibizumab 0.5mg — 0.5 mg ranibizumab (intravitreal injections) prefilled syringe)
  Other Names: Lucentis
  Arms: Group II ranibizumab 0.5 mg TER

SUMMARY:
This study was designed to evaluate the efficacy and safety of two different regimens of 0.5 mg ranibizumab given as intravitreal injection in patients with neovascular age-related macular degeneration

DETAILED DESCRIPTION:
This was a 12-month, phase IIIb, randomized, Visual Acuity assessor-masked, multi-center, interventional study assessing the efficacy and safety of the TER vs monthly regimens of 0.5 mg ranibizumab intravitreal (IVT) injections in patients with newly diagnosed nAMD. Patients will be randomized 1:1 into one of two treatment arms, Treat and Extend or monthly regimens.

There will be 3 periods in this study: Screening period (up to 14days), treatment period (11 months), follow-up period (1 month). At randomization visit patients will be randomized into one of the 2 treatment groups Group I ranibizumab 0.5 mg based on monthly treatment or Group II ranibizumab 0.5 mg based on TER (randomization ratio of 1:1) and will receive the first dose of Investigational treatment. Patients in Group I the following visits will perform on monthly intervals. For patients in Group II the investigator will evaluate disease activity (i.e., signs of exudation) based on SD-OCT, and in case of absence of disease activity every next visit will be 2 weeks), with a maximum of a 12-week interval.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients, ≥50 years of age with signed informed consent before study procedures
* Visual impairment predominantly due to nAMD.
* Active CNV secondary to AMD confirmed by presence of active leakage from CNV seen by fluorescein angiography (FA) and/or color fundus photography
* Presence of intra- or subretinal fluid/hemorrhage seen by SD-OCT
* BCVA score must be ≤ 78 and ≥ 23 letters at 4 meters starting distance using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity charts (approximate Snellen equivalent of 20/32 and 20/320)

Key Exclusion Criteria:

* Any type of advanced, severe or unstable disease, including any medical condition (controlled or uncontrolled) that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical status of the patient to a significant degree or put the patient at special risk.
* Stroke or myocardial infarction within 3 months prior to Screening.
* Any active periocular or ocular infection or inflammation in both eyes.
* Ocular disorders in the study eye at the time of enrollment that may confound interpretation of study results and compromise visual acuity.
* Presence of amblyopia or amaurosis in the fellow eye.
* History of treatment with any anti-angiogenic drugs (including any anti- vascular endothelial growth factor (anti-VEGF) agents) e.g., bevacizumab [Avastin®], aflibercept [Eylea®]) or vPDT in the study eye.
* History of intravitreal treatment with corticosteroids within 6 months and history of intra-ocular surgery within 3 months in the study eye prior to the Screening.
* Pregnant or nursing (lactating) women. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2015-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (80):
- Belgium (3):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Ottignies
  - Novartis Investigative Site, Zottegem
- Novartis Investigative Site, Santiago, Chile
- Novartis Investigative Site, Zagreb, Croatia, Croatia
- Denmark (2):
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Roskilde
- Egypt (2):
  - Novartis Investigative Site, Cairo, Abbassia
  - Novartis Investigative Site, Cairo
- Germany (15):
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Ahaus
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Siegburg
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Sulzbach
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Zalaegerszeg
- India (3):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Vanchiyoor, Thiruvanantapuram
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (7):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Udine, UD
- Portugal (4):
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Lisbon, Portugal
  - Novartis Investigative Site, Porto, Portugal
  - Novartis Investigative Site, Vila Franca de Xira, Portugal
- Russia (4):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Samara
- Slovakia (5):
  - Novartis Investigative Site, Banská Bystrica, Slovakia
  - Novartis Investigative Site, Nové Zámky, Slovakia
  - Novartis Investigative Site, Poprad, Slovakia
  - Novartis Investigative Site, Žilina, Slovakia
  - Novartis Investigative Site, Bratislava
- Novartis Investigative Site, Ljubljana, Slovenia, Slovenia
- South Korea (3):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
- Spain (6):
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Zaragoza, Zaragoza
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Ankara
- United Kingdom (8):
  - Novartis Investigative Site, Uxbridge, London
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Sunderland

REFERENCES:
- [Derived] Pawloff M, Bogunovic H, Gruber A, Michl M, Riedl S, Schmidt-Erfurth U. SYSTEMATIC CORRELATION OF CENTRAL SUBFIELD THICKNESS WITH RETINAL FLUID VOLUMES QUANTIFIED BY DEEP LEARNING IN THE MAJOR EXUDATIVE MACULAR DISEASES. Retina. 2022 May 1;42(5):831-841. doi: 10.1097/IAE.0000000000003385. PMID 34934034
- [Derived] Li E, Donati S, Lindsley KB, Krzystolik MG, Virgili G. Treatment regimens for administration of anti-vascular endothelial growth factor agents for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 May 5;5(5):CD012208. doi: 10.1002/14651858.CD012208.pub2. PMID 32374423
- [Derived] Waldstein SM, Coulibaly L, Riedl S, Sadeghipour A, Gerendas BS, Schmidt-Erfurth UM. Effect of posterior vitreous detachment on treat-and-extend versus monthly ranibizumab for neovascular age-related macular degeneration. Br J Ophthalmol. 2020 Jul;104(7):899-903. doi: 10.1136/bjophthalmol-2019-314661. Epub 2019 Sep 28. PMID 31563866

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized 1:1 into one of two treatment arms, Treat and Extend or monthly regimens.
  Safety set: One patient was randomized but did not receive at least one study treatment and did not record at least one post-baseline safety assessment
Groups:
- Group I Ranibizumab 0.5 mg TER: Ranibizumab 0.5 mg/0.05 mL (TER) treat and Extend regimen
- Group II Ranibizumab 0.5 mg Monthly: Ranibizumab 0.5 mg/0.05 mL (Monthly regimen)
Period: Overall Study
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Started | 323 | 327
Safety Set | 323 | 326
Completed | 290 | 295
Not Completed | 33 | 32
Not completed — Physician Decision | 1 | 3
Not completed — Protocol deviation | 1 | 2
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 14 | 17
Not completed — Adverse Event | 9 | 2
Not completed — Death | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly | Total
Number analyzed (Participants) | 323 | 327 | 650
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.3 (8.61) | 75.2 (8.13) | 75.2 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 181 | 360
  Male | 144 | 146 | 290

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline to Month 12
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. A positive average change from baseline of BCVA indicates improvement
Time Frame: Baseline to month 12
Population: The Full Analysis Set (FAS), comprised of all patients to whom treatment regimen had been assigned, was considered for the analysis. Only patients with the value for both Baseline and study completion after last observational carried forward (LOCF) were included in this analysis. LOCF was used as an imputation of missing data.
Measure: Least Squares Mean (Standard Error); unit: Letters (EDTRS)
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 320 | 323
Letters (EDTRS) | 6.2 (0.70) | 8.1 (0.70)
Statistical Analysis 1: Comparison: Group I Ranibizumab 0.5 mg TER vs Group II Ranibizumab 0.5 mg Monthly; Test type: Non-Inferiority or Equivalence — The following hypothesis was tested at a one-sided 0.025 level. Non-inferiority with respect to BCVA: H01: μtreat and extend - μmonthly ≤ - Δ versus HA1: μtreat and extend - μmonthly > - Δ where μtreat and extend and μmonthly are the unknown mean changes from baseline in BCVA to Month 12 in the treat and extend regimen and the monthly regimen, respectively. Δ is the non-inferiority margin and is pre-defined to be 5 letters for the justification of the margin; p < 0.001, ANCOVA

2. Secondary Outcome: Number of Visits Scheduled
Description: The number of visits scheduled according to the treat and extend regimen after treatment initiation
Time Frame: From Month1 to Month 11
Population: The Full Analysis Set (FAS), comprised of all patients to whom treatment regimen had been assigned, was analyzed.
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 323 | 327
Number of visits | 8.9 (2.56) | 11.2 (2.37)

3. Secondary Outcome: Change in BCVA From Baseline to Month 12
Description: Best Corrected Visual Acuity (BCVA) was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart at baseline and month 12 while participants were in a sitting position at a testing distance of 4 meters
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters (EDTRS)
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 320 | 323
Letters (EDTRS) | 6.4 (14.11) | 8.0 (11.61)

4. Secondary Outcome: Average BCVA Change From Baseline to Month 12
Description: Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters.
  Mean Visual Acuity was averaged over all monthly assessments from Baseline to Month 12
Time Frame: Baseline and every month for 12 months
Population: The Full Analysis Set (FAS), comprised of all patients to whom treatment regimen had been assigned, was considered for the analysis. Only patients with the value for both Baseline and average visual acuity (VA) from month 1 to study completion were included in this analysis.
Measure: Mean (Standard Deviation); unit: Letters (EDTRS)
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 320 | 323
Letters (EDTRS) | 6.3 (10.50) | 7.1 (9.41)

5. Secondary Outcome: Mean Change in Visual Acuity BCVA (Letters) From Baseline to Month 12
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) -like charts while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. For the mean change of best corrected visual acuity at Month 12 and compare to Baseline
Time Frame: Baseline and every month for 12 months
Population: The Full Analysis Set (FAS), comprised of all patients to whom treatment regimen had been assigned, was considered for the analysis. Only patients with the value for both Baseline and the specific post-baseline visit.
Measure: Mean (Standard Deviation); unit: Letters (EDTRS)
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 323 | 327
Letters (EDTRS)
  Month 1 (n=320, 322) | 4.6 (7.56) | 4.2 (6.98)
  Month 2 (n=240, 316) | 5.5 (8.64) | 5.8 (8.58)
  Month 3 (n=247, 311) | 6.7 (9.09) | 6.7 (9.19)
  Month 4 (n=213, 314) | 7.0 (10.90) | 7.3 (9.95)
  Month 5 (n=231, 302) | 6.0 (11.34) | 7.7 (10.61)
  month 6 (n=205, 302) | 6.9 (13.34) | 7.9 (10.83)
  Month 7 (n=230, 298) | 5.9 (14.25) | 7.9 (11.36)
  Month 8 (n=210, 295) | 7.5 (12.87) | 7.9 (11.34)
  Month 9 (n=179, 295) | 6.6 (13.63) | 7.6 (12.56)
  Month 10 (n=202, 296) | 6.3 (13.44) | 7.6 (12.06)
  Month 11 (n=180, 290) | 5.9 (14.12) | 7.5 (12.48)
  Month 12 (n=294, 295) | 6.6 (13.41) | 7.9 (11.96)

6. Secondary Outcome: Number of Patients With a BCVA Improvement of ≥1, ≥5, ≥10, ≥15, and ≥30 Letters From Baseline to Month 12
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An increased score indicates improvement in acuity. This outcome assessed the number of participants who had improvement of ≥1, ≥5, ≥10, ≥15, and ≥30 letters of visual acuity at Month 12 as compared with baseline
Time Frame: Baseline and every month for 12 months
Population: The Full Analysis Set (FAS), comprised of all patients to whom treatment regimen had been assigned, was considered for the analysis. Only patients with the value for both Baseline and the specific post-baseline visit were included for this analysis.
Measure: Number; unit: Number of participants
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 323 | 327
Number of participants
  Month 1,Gain of ≥ 1 letter (n=320,322) | 235 | 233
  Month 1, Gain of ≥ 5 letters | 145 | 145
  Month 1, Gain of ≥ 10 letters | 65 | 58
  Month 1, Gain of ≥ 15 letters | 24 | 23
  Month 1, Gain of ≥ 30 letters | 4 | 2
  Month 2, Gain of >= 1 letter (n=226, 316) | 168 | 244
  Month 2, Gain of >= 5 letters | 123 | 184
  Month 2, Gain of >= 10 letters | 60 | 88
  Month 2, Gain of >= 15 letters | 30 | 39
  Month 2, Gain of >= 30 letters | 4 | 3
  Month 3, Gain of >= 1 letter (n=161,311) | 120 | 244
  Month 3, Gain of >= 5 letters | 98 | 187
  Month 3, Gain of >= 10 letters | 57 | 110
  Month 3, Gain of >= 15 letters | 28 | 46
  Month 3, Gain of >= 30 letters | 2 | 3
  Month 4, Gain of >= 1 letter (n=128, 314) | 96 | 249
  Month 4, Gain of >= 5 letters | 67 | 198
  Month 4, Gain of >=10 letters | 48 | 118
  Month 4, Gain of >= 15 letters | 25 | 60
  Month 4, Gain of >= 30 letters | 4 | 8
  Month 5, Gain of >= 1 letter (n=114, 302) | 84 | 243
  Month 5, Gain of >= 5 letters | 64 | 197
  Month 5, Gain of >= 10 letters | 42 | 116
  Month 5, Gain of >= 15 letters | 19 | 59
  Month 5, Gain of >= 30 letters | 3 | 10
  Month 6, Gain of >= 1 letter (n=117, 302) | 85 | 238
  Month 6, Gain of >= 5 letters | 68 | 197
  Month 6, Gain of >= 10 letters | 42 | 125
  Month 6, Gain of >= 15 letters | 19 | 61
  Month 6, Gain of >= 30 letters | 2 | 11
  Month 7, Gain of >= 1 letter (n=176, 298) | 126 | 235
  Month 7, Gain of >= 5 letters | 94 | 196
  Month 7, Gain of >= 10 letters | 57 | 123
  Month 7, Gain of >= 15 letters | 33 | 69
  Month 7, Gain of >= 30 letters | 7 | 9
  Month 8, Gain of >= 1 letter (n=163, 295) | 124 | 228
  Month 8, Gain of >= 5 letters | 108 | 198
  Month 8, Gain of >= 10 letters | 69 | 130
  Month 8, Gain of >= 15 letters | 40 | 72
  Month 8, Gain of >= 30 letters | 4 | 9
  Month 9, Gain of >= 1 letter (n=129, 295) | 93 | 229
  Month 9, Gain of >= 5 letters | 78 | 186
  Month 9, Gain of >= 10 letters | 52 | 128
  Month 9, Gain of >= 15 letters | 28 | 70
  Month 9, Gain of >= 30 letters | 5 | 8
  Month 10, Gain of >= 1 letter (n=159, 296) | 113 | 230
  Month 10, Gain of >= 5 letters | 98 | 190
  Month 10, Gain of >= 10 letters | 60 | 126
  Month 10, Gain of >= 15 letters | 32 | 74
  Month 10, Gain of >= 30 letters | 4 | 10
  Month 11, Gain of >= 1 letter (131, 290) | 94 | 222
  Month 11, Gain of >= 5 letters | 79 | 187
  Month 11, Gain of >= 10 letters | 51 | 130
  Month 11, Gain of >= 15 letters | 32 | 74
  Month 11, Gain of >= 30 letters | 5 | 9
  Month 12, Gain of >= 1 letter (n=291, 295) | 217 | 226
  Month 12, Gain of >= 5 letters | 178 | 199
  Month 12, Gain of >= 10 letters | 123 | 135
  Month 12, Gain of >= 15 letters | 75 | 77
  Month 12, Gain of >= 30 letters | 12 | 8

7. Secondary Outcome: Number of Patients With Best Corrected Visual Acuity (BCVA) Loss <5, <10, and <15 Letters by Visit
Description: Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters.Best Corrected Visual Acuity (BCVA) was assessed in a sitting position using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters.
Time Frame: Baseline and every month for 12 months
Population: as for outcome 6
Measure: Number; unit: Number of participants
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 323 | 327
Number of participants
  Month 1, Loss of < 5 letters (n=320, 322) | 296 | 295
  Month 1, Loss of < 10 letters | 313 | 314
  Month 1, Loss of < 15 letters | 319 | 320
  Month 2, Loss of < 5 letters (n=226, 316) | 205 | 288
  Month 2, Loss of < 10 letters | 220 | 306
  Month 2, Loss of < 15 letters | 223 | 309
  Month 3, Loss of < 5 letters (n=161, 311) | 146 | 289
  Month 3, Loss of < 10 letters | 158 | 299
  Month 3, Loss of < 15 letters | 160 | 304
  Month 4, Loss of < 5 letters (n=128, 314) | 114 | 286
  Month 4, Loss of < 10 letters | 128 | 301
  Month 4, Loss of < 15 letters | 124 | 307
  Month 5, Loss of < 5 letters (n=114, 302) | 97 | 276
  Month 5, Loss of < 10 letters | 105 | 287
  Month 5, Loss of < 15 letters | 108 | 295
  Month 6, Loss of < 5 letters (n=117, 302) | 104 | 271
  Month 6, Loss of < 10 letters | 110 | 286
  Month 6, Loss of < 15 letters | 111 | 298
  Month 7, Loss of < 5 letters (n=176, 298) | 148 | 268
  Month 7, Loss of < 10 letters | 162 | 279
  Month 7, Loss of < 15 letters | 166 | 289
  Month 8, Loss of < 5 letters (n=163, 295) | 145 | 262
  Month 8, Loss of < 10 letters | 155 | 276
  Month 8, Loss of < 15 letters | 155 | 286
  Month 9, Loss of < 5 letters (n=129, 295) | 110 | 258
  Month 9, Loss of < 10 letters | 120 | 270
  Month 9, Loss of < 15 letters | 122 | 281
  Month 10, Loss of < 5 letters(n=159, 296) | 133 | 253
  Month 10, Loss of < 10 letters | 147 | 276
  Month 10, Loss of < 15 letters | 150 | 285
  Month 11, Loss of < 5 letters (n=131, 290) | 105 | 251
  Month 11, Loss of < 10 letters | 118 | 263
  Month 11, Loss of < 15 letters | 121 | 275
  Month 12, Loss of < 5 letters (291, 295) | 247 | 256
  Month 12, Loss of < 10 letters | 267 | 272
  Month 12, Loss of < 15 letters | 273 | 284

8. Secondary Outcome: Number of Patients With a BCVA Value of ≥ 73 Letters (Approximate 20/40 Snellen Chart Equivalent) at Month 12
Description: Best Corrected Visual Acuity (BCVA) was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts at baseline and month 12 while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. BCVA above 73 letters at Month 12 indicates a positive outcome
Time Frame: Baseline and every month for 12 months
Population: as for outcome 6
Measure: Number; unit: Number of participants
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 323 | 327
Number of participants
  Month 1 (n=320, 322) | 106 | 106
  Month 2 (n=226, 316) | 74 | 136
  Month 3 (n=161, 311) | 67 | 148
  Month 4 (n=128, 314) | 60 | 147
  Month 5 (n=114, 302) | 51 | 156
  Month 6 (n=117, 302) | 58 | 155
  Month 7 (n=176, 298) | 78 | 150
  Month 8 (n=163, 295) | 84 | 155
  Month 9 (n=129, 295) | 68 | 156
  Month 10 (n=159, 296) | 74 | 149
  Month 11 (n=131, 290 | 63 | 143
  Month 12 (n=291, 295) | 131 | 149

9. Secondary Outcome: The Mean Number of Treatment Frequency
Description: The number of injections received
Time Frame: Month 12
Population: Full Analysis Set (FAS) comprised all patients to whom treatment regimen had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment regimen they were assigned to at randomization
Measure: Mean (Standard Deviation); unit: Number of injections
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 323 | 327
Number of injections | 8.7 (2.68) | 11.0 (2.50)

10. Secondary Outcome: The Average Number of Days Between Injections
Description: The average dosing interval was measured as the average number of days between injections
Time Frame: Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 323 | 327
days | 40.3 (11.28) | 29.4 (3.27)

11. Secondary Outcome: Percentage of Participants With Fluid Free Macula Over Time up to Month 12
Description: OCT (optical coherence tomography) was used to assess intra-retinal fluid as Measured by SD-OCT (Spectral Domain-Optical Coherence Tomography). Fluid free macula refers to absence of macular edema (as assessed by the reading center). The full analysis set was used for this evaluation but the count presented are the counts of patients in the specific treatment group who have a value for the macular edema (center involvement) at study completion. These total counts are used as the denominator for the percentages
Time Frame: Month 12
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 291 | 290
Percentage of participants
  Absent | 60.5 | 60.7
  Definite | 39.5 | 39
  Can't grade | 0.0 | 0.3

12. Secondary Outcome: Change in Central Subfield Retinal Thickness (CSFT) Over Time
Description: OCT (optical coherence tomography) was used to assess CSFT (Central Sub-Field Thickness) representing the average retinal thickness of the circular area within 1 mm diameter around the foveal center. The Ns in the rows is the number of patients with a value for both baseline and the specific post-baseline visit
Time Frame: Month 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 323 | 327
microns
  Month 1 (n=311, 316) | -137.6 (132.33) | -126.8 (119.47)
  Month 2 (n=220, 311) | -151.6 (151.15) | -149.2 (137.60)
  Month 3 (n=157, 304) | -149.8 (167.26) | -151.8 (149.51)
  Month 4 (n=125, 307) | -141.8 (183.71) | -161.3 (149.36)
  Month 5 (n=110, 295) | -138.6 (160.04) | -160.9 (148.23)
  Month 6 (n=113, 298) | -140.1 (156.25) | -163.4 (157.18)
  Month 7 (n=173, 296) | -146.6 (160.72) | -166.9 (161.49)
  Month 8 (n=159, 290) | -153.4 (151.93) | -170.4 (156.68)
  Month 9 (n=126, 286) | -150.2 (153.82) | -169.3 (156.50)
  Month 10 (n=156, 291) | -154.6 (162.77) | -170.9 (153.90)
  Month 11 (n=127, 285) | -133.1 (170.47) | -174.8 (163.16)
  Month 12 (n=289, 287) | -172.1 (162.81) | -173.3 (154.13)

13. Secondary Outcome: Percentage of Patients With Choroidal Neovascularization (CNV) Leakage Assessed by Fluorescein Angiography (FA) in the Study Eye at
Description: To evaluate presence of active CNV leakage on fluorescein angiography (FA) by reading center over time up to Month 12. The full analysis set was used for this evaluation but the count presented are the counts of patients in the specific treatment group who have a value for the presence of leakage at study completion. These total counts are used as the denominator for the percentages.
Time Frame: Month 12
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 278 | 286
Percentage of participants
  Yes | 18.7 | 17.1
  No | 74.1 | 76.9
  Can't grade | 0.0 | 2.4
  Not applicable | 7.2 | 3.5

14. Secondary Outcome: Change From Baseline in Composite Score of the National Eye Institute-Visual Function Questionnaire-25 (NEI-VFQ-25)
Description: The survey consisted of 25 items representing 11 vision related constructs (general vision, ocular pain, near activities, distance activities, social functioning, mental health, role difficulties, dependency, driving, color vision, peripheral vision) plus a single-item general health rating question. The score of each individual question ranged from 0 (worst) to 100 which indicates the best possible response. The composite score and score of each of each construct also ranged from 0 to 100 as they are calculated as total scores divided by the number of questions. The higher the values of total scores represent better outcome
Time Frame: Baseline, Month 12
Population: The Full Analysis Set (FAS), comprised of all patients to whom treatment regimen had been assigned, was considered for the analysis. Only patients with the value for both Baseline and post-baseline value at the specific visit were included for this analysis
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Number analyzed (Participants) | 290 | 293
Score on a scale | 2.3 (13.93) | 4 (13.72)

ADVERSE EVENTS:
Arm/Group | Group I Ranibizumab 0.5 mg TER | Group II Ranibizumab 0.5 mg Monthly
Serious Adverse Events (participants affected / at risk) | 39/323 | 42/326
Other Adverse Events (participants affected / at risk) | 164/323 | 166/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I Ranibizumab 0.5 mg TER (N=323) | Group II Ranibizumab 0.5 mg Monthly (N=326)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Cataract (Fellow eye) (Eye disorders) | 1 | 0
Corneal erosion (Study eye) (Eye disorders) | 1 | 0
Corneal infiltrates (Study eye) (Eye disorders) | 1 | 0
Dacryostenosis acquired (Fellow eye) (Eye disorders) | 0 | 1
Dacryostenosis acquired (Study eye) (Eye disorders) | 0 | 1
Macular hole (Study eye) (Eye disorders) | 0 | 1
Retinal detachment (Study eye) (Eye disorders) | 1 | 0
Retinal haemorrhage (Study eye) (Eye disorders) | 1 | 0
Retinal tear (Study eye) (Eye disorders) | 1 | 0
Vitreous haemorrhage (Study eye) (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Endophthalmitis (Fellow eye) (Infections and infestations) | 0 | 1
Endophthalmitis (Study eye) (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 2
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1
Intraocular pressure increased (Fellow eye) (Investigations) | 0 | 1
Intraocular pressure increased (Study eye) (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 3 | 1
VIth nerve paresis (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I Ranibizumab 0.5 mg TER (N=323) | Group II Ranibizumab 0.5 mg Monthly (N=326)
Age-related macular degeneration (Fellow eye) (Eye disorders) | 9 | 4
Blepharitis (Fellow eye) (Eye disorders) | 6 | 8
Blepharitis (Study eye) (Eye disorders) | 5 | 6
Cataract (Fellow eye) (Eye disorders) | 7 | 10
Cataract (Study eye) (Eye disorders) | 7 | 7
Choroidal neovascularisation (Fellow eye) (Eye disorders) | 6 | 7
Conjunctival haemorrhage (Study eye) (Eye disorders) | 14 | 19
Detachment of retinal pigment epithelium (Study eye) (Eye disorders) | 0 | 4
Dry eye (Fellow eye) (Eye disorders) | 7 | 6
Dry eye (Study eye) (Eye disorders) | 6 | 7
Eye pain (Study eye) (Eye disorders) | 10 | 5
Neovascular age-related macular degeneration (Fellow eye) (Eye disorders) | 8 | 16
Ocular hypertension (Study eye) (Eye disorders) | 4 | 4
Punctate keratitis (Study eye) (Eye disorders) | 4 | 3
Retinal haemorrhage (Study eye) (Eye disorders) | 5 | 8
Retinal pigment epithelial tear (Study eye) (Eye disorders) | 4 | 3
Visual acuity reduced (Fellow eye) (Eye disorders) | 6 | 4
Visual acuity reduced (Study eye) (Eye disorders) | 15 | 12
Vitreous floaters (Study eye) (Eye disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 4 | 5
Oedema peripheral (General disorders) | 0 | 5
Bronchitis (Infections and infestations) | 6 | 12
Conjunctivitis (Fellow eye) (Infections and infestations) | 6 | 6
Conjunctivitis (Study eye) (Infections and infestations) | 10 | 6
Cystitis (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 9 | 12
Nasopharyngitis (Infections and infestations) | 18 | 26
Respiratory tract infection (Infections and infestations) | 5 | 3
Sinusitis (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 5 | 2
Blood pressure increased (Investigations) | 4 | 1
Intraocular pressure increased (Fellow eye) (Investigations) | 3 | 8
Intraocular pressure increased (Study eye) (Investigations) | 27 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Dizziness (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 4 | 4
Sciatica (Nervous system disorders) | 6 | 1
Depression (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 5 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Hypertension (Vascular disorders) | 23 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety